CLINICAL TRIAL: NCT01009112
Title: Treating Insomnia & Nightmares After Trauma: Impact on Symptoms & Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Sean P.A. Drummond, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1RC1NR011728-01 (NIH)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Nightmares; Insomnia; Posttraumatic Stress Disorder
Keywords: Sleep; Sleep Disorder; Veterans; Active Duty; OEF; OIF; PTSD
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic; Sleep Wake Disorders | interventions — Implosive Therapy; Cognitive Behavioral Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CBT for Insomnia (Experimental): Patients change their sleep times and habits in order to reduce alertness and "over thinking" when they are trying to sleep. This helps them learn how to sleep overnight in one solid block of time
  Interventions: Behavioral: PTSD + IRT/CBT-I
- Imagery Rehearsal Therapy (Experimental): Patients "rescript" the narrative of a nightmare to eliminate the distressing elements and create a new pleasant dream scene. They then rehearse this scene in their imagination at least twice each day. This reduces the frequency and intensity of the target nightmare and often reduces other nightmares, too.
  Interventions: Behavioral: PTSD + IRT/CBT-I
- Prolonged Exposure (Experimental): This behavioral treatment for PTSD involves 1) systematic and repeated exposure to objects and situations that are avoided due to trauma-related distress, 2) prolonged, repeated recounting of trauma memories through visualization, and 3)therapist-guided discussions of thoughts and emotions related to the exposure exercises. The goals of PE are to reduce the anxiety and distress elicited by trauma-related memories and situations, show patients these memories and situations are distinct from the trauma, and teach patients they can tolerate the distress caused by these memories and situations.
  Interventions: Behavioral: PTSD + IRT/CBT-I; Behavioral: PTSD + Supportive Care Therapy
- Suportive Care Therapy (Active Comparator): This is an active therapy where the focus of the intervention is on helping patients better understand their emotional response to their PTSD and sleep symptoms.
  Interventions: Behavioral: PTSD + Supportive Care Therapy

INTERVENTIONS:
Behavioral: PTSD + IRT/CBT-I — 6 weeks of prolonged exposure, 5 weeks of imagery rehearsal therapy, and 7 weeks of cognitive behavioral therapy for insomnia
  Other Names: IRT; PE; exposure therapy; Cognitive Behavioral Therapy for Insomnia
  Arms: CBT for Insomnia; Imagery Rehearsal Therapy; Prolonged Exposure
Behavioral: PTSD + Supportive Care Therapy — 6 weeks of prolonged exposure + 12 weeks of supportive care therapy
  Other Names: PE; exposure therapy
  Arms: Prolonged Exposure; Suportive Care Therapy

SUMMARY:
Exposure to trauma, especially when it manifests as Posttraumatic Stress Disorder (PTSD), results in numerous negative consequences for patients, families, and society. Some of the most frequent, disturbing, and treatment resistant symptoms of PTSD are nightmares and insomnia. This study will examine whether treatments specifically targeted at those sleep disorders can improve clinical outcomes and increase health-related quality of life in individuals recently exposed to war-related trauma. Hypotheses are that treating nightmares and insomnia will improve both nighttime and daytime symptoms of PTSD, as well as quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 1 or more deployments to OEF or OIF
* Exposure to Trauma
* Nightmares 2 or more times per week
* Insomnia for 1 month or more
* Live in greater San Diego County region

Exclusion Criteria:

* Use of medications for sleep or nightmares in the past 2 weeks
* Current enrollment in psychotherapy for PTSD
* Current or recent substance or alcohol abuse or dependence
* Other untreated sleep disorders (e.g., sleep apnea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
nightmares and insomnia symptoms | pre-treatment; weeks 6, 11, and 18 of treatment; 3-month follow-up post-treatment

SECONDARY OUTCOMES:
daytime (non-sleep) PTSD symptoms | pre-treatment; weeks 6, 11, and 18 of treatment; 3-month follow-up post-treatment
health-related quality of life | pre-treatment; weeks 6, 11, and 18 of treatment; 3-month follow-up post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sean PA Drummond, PhD, Principal Investigator — Veterans Medical Research Foundation & University of California San Diego
Locations (1):
- Veterans Affairs San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Derived] Mascaro L, Phillips AJK, Clark JW, Straus LD, Drummond SPA. Diurnal Rhythm Robustness in Individuals With PTSD and Insomnia and The Association With Sleep. J Biol Rhythms. 2021 Apr;36(2):185-195. doi: 10.1177/0748730420984563. Epub 2021 Jan 20. PMID 33472513
- [Derived] Walters EM, Jenkins MM, Nappi CM, Clark J, Lies J, Norman SB, Drummond SPA. The impact of prolonged exposure on sleep and enhancing treatment outcomes with evidence-based sleep interventions: A pilot study. Psychol Trauma. 2020 Feb;12(2):175-185. doi: 10.1037/tra0000478. Epub 2019 Jun 27. PMID 31246050